CLINICAL TRIAL: NCT05273879
Title: Necessity of Fusion Following Decompression Surgery in Patients With Single-level Lumbar Stenosis: Study Protocol for an Open-label Multicenter Non-inferiority Randomized Controlled Clinical Trial
Brief Title: Necessity of Fusion Following Decompression Surgery in Patients With Single-level Lumbar Stenosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sklifosovsky Institute of Emergency Care (Other Government)
Collaborators: Pirogov National Medical Surgical Center (Other Government); Moscow Scientific and Practical Center of Medical Rehabilitation, Restorative and Sports Medicine (Other)
Responsible Party: Principal Investigator, Ivan Lvov, MD, PhD, Senior fellow, Sklifosovsky Institute of Emergency Care
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03\2022
Record Dates: First submitted 2022-02-19; First posted 2022-03-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Lumbar Spinal Stenosis; Spinal Stenosis; Spinal Fusion
Keywords: lumbar spine; lumbar fusion; laminotomy; decompression without fusion; lumbar stenosis
MeSH Terms: conditions — Spinal Stenosis; Constriction, Pathologic | interventions — Decompression; Gene Fusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- decompression group (Other): minimally invasive decompression without fusion
  Interventions: Procedure: decompression
- fusion group (Other): minimally invasive decompression with trans-foraminal interbody fusion
  Interventions: Procedure: fusion

INTERVENTIONS:
Procedure: decompression — laminotomy of the corresponding adjacent vertebrae, partial flavectomy and medial facetectomy are planned to be performed unilaterally. Depending on the surgeon's personal preferences, the following two options are available: 1) equivalent decompression procedure contralaterally and 2) crossover contralateral decompression. Irrespective of the selected option, the spinous process, the interspinous and supraspinous ligaments, part of the facet joints, and the corresponding part of the vertebral arch must be preserved intact in all participants.
  Arms: decompression group
Procedure: fusion — First, decompression is performed according to one of the above methods. Next, trans-foraminal interbody fusion with a cage (TLIF) and fixation with pedicle screws are performed.
  Arms: fusion group

SUMMARY:
Long-term clinical results of two methods of surgical treatment (spinal decompression with or without fusion) in patients with single-level lumbar stenosis will be compared. A clear framework for surgical treatment methods and standardized postoperative rehabilitation treatment will be set to obtain the maximum homogeneity of the patient groups.

This trial should provide the first level of evidence for the need for spinal fusion in patients with single-level lumbar stenosis, subject to the high homogeneous comparison groups. Additional results will allow comparing the economic aspects of different surgical treatments for 2 years after surgery.

DETAILED DESCRIPTION:
The necessity of spinal segment fusion after decompression is one of the most controversial and unresolved issues in single-level lumbar spinal stenosis surgery. To date, only one trial carried out 15 years ago focused on this problem. The key purpose of the current trial is to compare the long-term clinical results of the two surgical methods (decompression vs. decompression and fusion) in patients with single-level lumbar stenosis.

This study is focused on the non-inferior clinical results of decompression compared with the standard fusion procedure. In the decompression group, the spinous process, the interspinous and supraspinous ligaments, part of the facet joints, and corresponding parts of the vertebral arch are to be preserved intact. In the fusion group, decompression is to be supplemented with transforaminal interbody fusion. Participants meeting the inclusion criteria will be randomly divided into two equal groups (1:1), depending on the surgical method. The final analysis will include 86 patients (43 per group). The primary endpoint is Oswestry Disability Index dynamics at the end of the 24-month follow-up compared to the baseline level. Secondary outcomes included those estimated using the SF-36 scale, EQ-5D-5L, and psychological scales. Additional parameters will include sagittal balance of the spine, fusion results, total cost of surgery, and hospital stay followed by two-year treatment. Follow-up examinations will be performed at 3, 6, 12, and 24 months Authors suggest that this study will improve the evidence for application of various surgical techniques for lumbar spine stenosis surgery and verify the existing protocol for surgical management.

ELIGIBILITY:
Inclusion Criteria:

* age of patients from 45 to 75 years;
* stenosis C or D according to Shizas et al. according to MRI at the level of L2-L3, L3-L4, L4-L5 or L5-S1;
* clinical manifestations of lumbar stenosis (neurogenic claudication syndrome and/or radiculopathy);
* lack of effect from conservative therapy within 3 months;
* Informed consent to take part in the study.

Exclusion Criteria:

* spondylolisthesis more than 3 mm;
* spinal instability according to functional radiography;
* sagittal imbalance (type 4 according to C. Barrey);
* bone density of the vertebrae at the level of the operation is less than 100 HU;
* clinically significant spinal stenosis at 2 or more levels;
* previously performed surgeries on the spine;
* risk of anesthesia 4 or 5 according to ASA;
* inability to take part in control examinations within 2 years after the operation;
* participation in other clinical trials related to surgical or conservative treatment of diseases of the spine.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index | 24 months
  The questionnaire includes 10 sections containing 6 statements each. Depending on the answer, a score is assigned (from 0 to 5). The maximum number of points is 50. After that, the points are converted into percentages (from 0 to 100%).

SECONDARY OUTCOMES:
SF-36 v.1 scale (standard form) | 24 months
  The questionnaire contains 36 questions, grouped into 8 scales that assess physical functioning, role-playing, bodily pain, general health, vitality, social functioning, emotional state, and mental health. For each of them, the maximum score is 100 points.
EQ-5D-5L | 24 months
  The questionnaire contains 5 sections (mobility, self-care, usual activities, pain, anxiety) of three statements and the EQ-VAS visual analog pain scale. The results can be converted into a single numerical value (index) adjusted for the patient's region of residence
Won-Korff Chronic Pain Syndrome Assessment Scale | 24 months
  allows evaluating the severity of pain and its impact on life in points. Grade 0 corresponds to the absence of pain, and grade IV to the maximum limitation of life because of severe pain.
Pain Catastrophizing Scale | 24 months
  makes it possible to assess completely the psychological aspects of pain perception, in particular the exaggerated negative perception of painful stimuli. The questionnaire contains 13 questions, each of which is evaluated in points (0 points, no symptom, 4, the patient experiences these feelings all the time).
Chronic Pain Coping Inventory | 24 months
  allow one of eight scales to classify a patient's preferred strategy for coping with chronic pain.
scale of the American Society of Anesthesiologists ASA | baseline
  This classification distinguishes 5 classes of physical status depending on the presence of concomitant diseases (Class I, healthy patient, Class V, dying).
The cost of the treatment | 24 months
  The cost of hospitalization of the patient, including the performance of surgical intervention, as well as the period of the patient's incapacity for work because of spinal disease, will also be calculated. Also, within 2 years after the intervention, the cost of subsequent treatment in rehabilitation centers and other hospitals for complications of the operation or other manifestations of degenerative-dystrophic changes in the lumbar spine will be considered.
quality of fusion | 24 months
  according to CT data, the quality of fusion using the Tan criteria will be graded into one of four grades of fusion-grade I (complete fusion) to grade IV (bipolar pseudarthrosis)
pelvic tilt (PT) | 24 months
  a parameter defined as the angle created by a line running from the sacral endplate midpoint to the center of the bifemoral heads and the vertical axis. Will be evaluated on X-ray.
pelvic incidence (PI) | 24 months
  the angle between the line perpendicular to the sacral endplate at its midpoint and a line connecting this point to the axis of the femoral head. Will be evaluated on X-ray.
sacral slope (SS) | 24 months
  the angle between the tangent line to the superior endplate of S1 and the horizontal plane. Will be evaluated on X-ray.
al axis displacement (SVA) | 24 months
  a horizontal distance between a plumb line dropped from the center of the C7 body and the posterior-superior corner of the S1 body. Will be evaluated on X-ray.

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Grin, MD, PhD, Study Chair — Sklifosovsky Research Institute for Emergency Medicine
Locations (2):
- Russia (2):
  - Pirogov National Medical and Surgical Center, Moscow, Moscow
  - Sklifosovsky Research Institute for Emergency Medicine, Moscow, Moscow

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request in Sklifosovsky Research Institute for Emergency Medicine
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Study protocol will be available after march 2022. An interim analysis will be conducted when follow-up data is available at 12 months for at least 20 patients in each cohort. Final analysis will be presented after december 2026
Access Criteria: the approval of institutional review board

REFERENCES:
- [Derived] Grin A, Lvov I, Talypov A, Smirnov V, Kordonskiy A, Lebedev V, Zuev A, Senko I, Pogonchenkova I, Krylov V. Necessity of fusion following decompression surgery in patients with single-level lumbar stenosis: study protocol for an open-label multicentre non-inferiority randomized controlled clinical trial. Trials. 2023 Jul 10;24(1):451. doi: 10.1186/s13063-023-07486-8. PMID 37430281